CLINICAL TRIAL: NCT06287918
Title: A First-in-human, Open-label, Dose Escalation and Expansion Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Activity of 3HP-2827 in Patients With Unresectable or Metastatic Solid Tumors With FGFR2 Alterations
Brief Title: A First-in-human Study of 3HP-2827 in Patients With Unresectable or Metastatic Solid Tumors With FGFR2 Alterations
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: 3H (Suzhou) Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3HP-2827-101
Record Dates: First submitted 2024-02-22; First posted 2024-03-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors With FGFR2 Alterations, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stage I - dose escalation (Experimental): Dose escalation of 3HP-2827 in patients with advanced solid tumors.
  Interventions: Drug: 3HP-2827
- Stage II - expansion (Experimental): Expansion evaluating the recommended dose and schedule of 3HP-2827 identified from Stage I.
  Interventions: Drug: 3HP-2827

INTERVENTIONS:
Drug: 3HP-2827 — 3HP-2827 will be administered orally once daily in 28-day cycles.

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of 3HP-2827 in the treatment of unresectable or metastatic solid tumors with FGFR2 alterations. Patients will be enrolled in two stages: dose escalation stage (Stage I) and expansion stage (Stage II).

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and able to provide written informed consent and has the ability to comply with the study protocol
* Men or women, age ≥ 18 years at the time of signing informed consent.
* Histologically or cytologically confirmed surgically unresectable, locally advanced, metastatic solid tumor.
* ECOG score is 0 or 1.
* An expected survival of ≥ 12 weeks.
* Evaluable or measurable disease per RECIST v1.1.
* Adequate organ function, as measured by laboratory values.

Exclusion Criteria:

* Active brain metastases.
* Have other malignancies within the past 3 years.
* The toxicity from previous anti-tumor treatment has not recovered to ≤ grade 1.
* Clinically significant corneal or retinal disease/keratopathy.
* Clinically significant cardiovascular disorders.
* Failure to swallow, chronic diarrhea, or presence of other factors affecting drug absorption.
* Known to be allergic to any study drug or any of its excipients.
* Any other diseases or clinical laboratory, etc that may affect the interpretation of the results, or renders the patients at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Stage- incidence of adverse events (AEs) | From baseline up until 28 days after the final dose
Dose Escalation Stage- incidence of dose-limiting toxicities (DLTs) | Days 1-28 of Cycle 1 (a cycle is 28 days)
Dose Escalation Stage -Percentage of Participants With Changes From Baseline in Targeted Vital Signs | From baseline up until 28 days after the final dose
Dose Escalation Stage -Percentage of Participants With Changes From Baseline in Targeted Clinical Laboratory Test Results | From baseline up until 28 days after the final dose
Dose Escalation Stage -Percentage of Participants With Changes From Baseline in Targeted ECG Parameters | From baseline up until 28 days after the final dose
Dose Escalation Stage -determine the maximum tolerated dose (MTD) and/or the recommended dose (RD) for expansion stage or recommended Phase II dose (RP2D) of 3HP-2827 | Initiation of study drug until study discontinuation, (up to approximately 24 months)
Expansion stage -Objective response rate（ORR） | Initiation of study drug until disease progression (up to approximately 36 months)

SECONDARY OUTCOMES:
Plasma Concentration of 3HP-2827 and/or its major metabolites | Initiation of study drug until study discontinuation（up to 45 months）
Duration of Response (DOR) as assessed by RECIST v1.1 | Up to 45 months
Progression-free survival (PFS) as assessed by RECIST v1.1 | Up to 45 months
Overall survival | Up to 48 months
Dose escalation stage - Objective Response Rate (ORR) | Up to 45 months
Expansion Stage- incidence of adverse events (AEs) | From baseline up until 28 days after the final dose
Expansion Stage -Percentage of Participants With Changes From Baseline in Targeted Vital Signs | From baseline up until 28 days after the final dose
Expansion Stage -Percentage of Participants With Changes From Baseline in Targeted Clinical Laboratory Test Results | From baseline up until 28 days after the final dose
Expansion Stage -Percentage of Participants With Changes From Baseline in Targeted ECG Parameters | From baseline up until 28 days after the final dose

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic, Phoenix, Arizona
  - The University of Texas MD Anderson Cancer Center, Houston, Texas